CLINICAL TRIAL: NCT05905705
Title: Disruptions of Brain Networks and Sleep by Electroconvulsive Therapy
Acronym: DNS-ECT
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, MohammadMehdi Kafashan, Instructor, Washington University School of Medicine
Other Study IDs: 202204161; K01MH128663 (NIH)
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Electroencephalography (EEG) — High-density EEG will be acquired during resting wakefulness before each ECT session.
Diagnostic Test: Quantitative Measurements of Sleep Microstructure — Overnight sleep EEG will be recorded one day before each ECT session using the DREEM device. The DREEM device allows continuous recording of multichannel EEG.

SUMMARY:
Electroconvulsive therapy (ECT) alleviates treatment-resistant depression (TRD) through repeated generalized seizures. The goal of this study is to evaluate how ECT impacts sleep-wake regulation and efficiency of information transfer in functional networks in different states of arousal.

DETAILED DESCRIPTION:
Graph-based network analyses of electroencephalographic (EEG) signals allow characterization of functional networks. The robustness of local networks to disruption is quantified as local efficiency (Elocal), while network integration is quantified as global information transfer (Eglobal).

Aim 1: Assess relationships between sleep slow-wave activity (SWA) and awake Elocal over the course of ECT.

Aim 2: Quantify relationships between depression severity and awake Elocal over the course of ECT.

ELIGIBILITY:
Inclusion Criteria:

* Referral for initial ECT index course for Treatment-Resistant Depression (TRD), unipolar major depressive disorder or bipolar depression. Historic failure of response or remission to at least two antidepressant medications of sufficient dose and duration will be used for TRD diagnostic.

Exclusion Criteria:

* Diagnoses of schizophrenia or schizoaffective disorders.
* Subjects who are unable to tolerate the Dreem device for sleep recordings will be excluded from the study.

Ages: 21 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Treatment-Resistant Depression (TRD), unipolar major depressive disorder or bipolar depression
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Slow wave activity (SWA) during non-rapid eye movement sleep (NREM) stage N2/N3 | Up to 4 weeks during patients ECT treatment course
  Total power of EEG slow waves per minute present during N2/N3 sleep
Graph-based neural connectivity measure of local efficiency of information transfer (Elocal) during wakefulness | Up to 4 weeks during patients ECT treatment course
  Elocal will be calculated as the average inverse shortest path length among neighbors of a node within the network. Nodes will be constructed based on 5-minute recordings of eyes closed wakefulness theta band (4-8 Hz) EEG.
Graph-based neural connectivity measure of global information transfer (Eglobal) during ECT-induced seizure | Up to 4 weeks during patients ECT treatment course
  Eglobal will be calculated as the average inverse shortest path length between node pairs in the networks. Nodes will be constructed based on ECT-induced seizure EEG data within the alpha band (8-13 Hz).

CONTACTS AND LOCATIONS:
Overall Officials: MohammadMehdi Kafashan, Principal Investigator — Washington University School of Medicine in St. Louis
Locations (1):
- Washington University School of Medicine/Barnes-Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Subramanian S, Labonte AK, Nguyen T, Luong AH, Hyche O, Smith SK, Hogan RE, Farber NB, Palanca BJA, Kafashan M; CET-REM Study Group. Correlating electroconvulsive therapy response to electroencephalographic markers: Study protocol. Front Psychiatry. 2022 Nov 3;13:996733. doi: 10.3389/fpsyt.2022.996733. eCollection 2022. PMID 36405897
- [Background] Hill AT, Zomorrodi R, Hadas I, Farzan F, Voineskos D, Throop A, Fitzgerald PB, Blumberger DM, Daskalakis ZJ. Resting-state electroencephalographic functional network alterations in major depressive disorder following magnetic seizure therapy. Prog Neuropsychopharmacol Biol Psychiatry. 2021 Jun 8;108:110082. doi: 10.1016/j.pnpbp.2020.110082. Epub 2020 Aug 24. PMID 32853716
- [Derived] Kafashan M, Lebovitz L, Greenspan R, Zhao S, Kim T, Husain M, Hershey T, Cristancho P, Hogan RE, Palanca BJA, Farber NB; DNS-ECT Study Team. Investigating the impact of electroconvulsive therapy on brain networks and sleep: an observational study protocol. BMJ Open. 2025 Mar 7;15(3):e098859. doi: 10.1136/bmjopen-2025-098859. PMID 40054874